CLINICAL TRIAL: NCT01887873
Title: An Open Two-center Study Evaluating the Safety of Hyaluronan Thiomer i.o. Implant During Combined Phacoemulsification - Non Penetrating Deep Sclerectomy in Patients With Open Angle Glaucoma and Cataract
Brief Title: Safety of Hyaluronan Thiomer i.o. Implant During Combined Phacoemulsification - Non Penetrating Deep Sclerectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPHT150611
Record Dates: First submitted 2013-06-11; First posted 2013-06-27 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2013-06

CONDITIONS: Open Angle Glaucoma; Cataract
Keywords: open angle glaucoma; cataract
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyaluronan Thiomer i.o. implantable device (Other): active treatment
  Interventions: Device: Hyaluronan Thiomer i.o. implant

INTERVENTIONS:
Device: Hyaluronan Thiomer i.o. implant

SUMMARY:
The study is designed to assess the safety of Hyaluronan Thiomer i.o. implant in patients with primary open angle glaucoma undergoing a combined phacoemulsification - non penetrating deep sclerectomy procedure.

In this study, Hyaluronan Thiomer i.o. will be implanted during a combined surgery of cataract and non - penetrating deep sclerectomy in a group of 16 patients with primary open angle glaucoma and clinically significant cataract. Given that a considerable number of glaucoma patients also suffer from cataract, it is reasonable to test Hyaluronan Thiomer i.o. during a combined procedure of phacoemulsification and deep sclerectomy. This is also of importance because a combined procedure avoids the need of a second operation in this group of patients. Finally, it has been shown that combined phacoemulsification - deep sclerectomy does not induce a further risk compared to deep sclerectomy alone(open phase I study).

Safety will be assessed based on the occurrence of adverse events.

Efficacy assessments will be performed at every visit and efficacy analysis will include:

* Proportion of subjects at each study time point which will need additional IOP lowering drug therapy to achieve an IOP reduction to values < 21 mmHg. If a subject needs more than one drug to achieve target IOP, the number of drugs needed to achieve adequate IOP reduction will be recorded.
* Proportion of subjects at each time point which will need Neodymium:YAG goniopuncture to achieve an IOP reduction to values < 21 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Primary open angle glaucoma with uncontrolled IOP (IOP > 21 mmHg or more) despite maximally tolerated topical medication
* Clinically significant cataract as judged by the investigator
* Scheduled for combined cataract/glaucoma surgery

Exclusion Criteria:

Any of the following will exclude a subject from the study:

* Participation in a clinical trial in the 3 weeks preceding the study
* Presence or history of a severe medical condition as judged by the clinical investigator
* Wearing of contact lenses
* Loss of mean deviation of visual field testing of 15 dB or more
* Diabetic retinopathy
* Dysgenetic glaucoma, secondary glaucoma or any type of angle closure glaucoma
* Previous argon laser trabeculoplasty
* Severe dry eye syndrome as judged by the investigator
* Ocular infection or clinically significant inflammation as judged by the investigator
* Ocular surgery in the 12 months preceding the study
* History of glaucoma surgery in the study eye
* Neovascular form of age related macular degeneration
* The following lenses will not be implanted during cataract surgery Multifocal lenses Toric lenses PMMA lenses
* Ametropy >/= 6 Dpt
* Patients in which the surgical procedure cannot be performed or completed according to the protocol for any reason will be excluded and replaced.
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety | Safety will be assessed up to 12 months.
  Safety will be based on the occurrence of adverse events.

SECONDARY OUTCOMES:
Efficacy | Efficacy assessments will be performed up to 12 months.
  Efficacy will be assessed based on postoperative IOP reduction, assessment of the proportion of subjects needing additional IOP lowering medication and the proportion of subjects needing postoperative Neodymium:YAG goniopuncture.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Medical University of Vienna, Austria, Vienna, Austria